CLINICAL TRIAL: NCT05072301
Title: Preliminary Test of Reactive Carrot Incentives in a Practice Quit Environment With Contingency Management Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000030430
Record Dates: First submitted 2021-09-30; First posted 2021-10-08 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation
Keywords: incentives
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): The treatment group will receive a onetime offer of $80 (a reactive carrot) to forego all abstinence (contingency management) reward payments in the future.
  Interventions: Behavioral: Contingency Management
- Control (Placebo Comparator): The control group will receive contingency management payments and other monetary benefits for completing the trial.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Contingency Management — The treatment group will receive a onetime offer of $80 (a reactive carrot) to forego all abstinence (contingency management) reward payments in the future.
  Arms: Contingency Management
Behavioral: Control — The control group will receive contingency management payments and other monetary benefits for completing the trial.
  Arms: Control

SUMMARY:
The primary aim of this study is to pilot test a novel reactive carrot approach for improving individuals' ability to stick to a "practice quit" program in a smoking cessation context. In this study, the treatment gives subjects an offer to forego a monetary incentive to forego the opportunity to receive subsequent abstention (contingency management) rewards.

DETAILED DESCRIPTION:
All the subjects, treatment and control groups, would be given the opportunity to receive attendance rewards for attending six CO testing meetings as well as abstention (contingency management) rewards for abstaining from smoking. The only difference between the subjects randomly assigned to treatment and control groups is that each member of the treatment group would be tempted at the beginning of their program by being offered a one-time monetary incentive to forego the opportunity to receive subsequent abstention (contingency management) rewards. Treatment group subjects would, at their initial intake meeting after the attendance and abstention rewards opportunity had been described, be given a one-time opportunity to received $80 temptation payment to give up the opportunity to receive subsequent abstinence (contingency management) rewards that could be worth as much as $165. Subjects who accepted this one-time opportunity would remain enrolled in the practice quit smoking and they would still be eligible to receive attendance reward compensation totaling up to $30 for showing up to their six testing appointments. The purpose of the study is to test whether resisting the temptation to accept the one-time payment helps steel the resolve of the treatment subjects to follow through and make sure that they earn the subsequent contingency management rewards. More specifically, an intent-to-treat design will allow us to test whether the temptation causes treatment group subjects to have greater success than the un-tempted control group subjects to abstain from smoking during the two-week practice quit period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Smoke ≥ 3 cigarettes per week and expressing interest in quitting smoking.

Exclusion Criteria:

* Unstable psychiatric conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia
* unstable medical conditions that have not been well controlled (e.g., acute infection requiring hospitalization) for the past 30 days
* pregnant or breastfeeding women
* those with limited decision making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Breath Carbon Monoxide Test (measured in ppm levels) | 14 days following intake date
  A primary outcome is the sum of times a subject tested abstinent at the 6 CO testing meetings. To test for abstinence, a breath carbon monoxide test will be used to determine exposure to smoke. Abstinence will be coded as expired-air carbon monoxide (CO) levels below 5 ppm.
Proportion of CO (CO ≤ 4ppm) | 14 days following intake date
  Proportion of 6 CO tests showing abstinence (CO ≤ 4ppm)
Maximum number of consecutive abstinent days | 14 days following intake date
  The maximum number of consecutive abstinent days for each subject will be measured

SECONDARY OUTCOMES:
Attrition | 14 days following intake date
  Attrition will be measured by participants ability to make their testing appointments.
Contingency Management Payment | 14 days following intake date
  Total amount of abstention (contingency management) rewards paid to subjects.
Time to first relapse | 14 days following intake date
  Time to first relapse will be measured by subjects self-reporting use of different types of tobacco products or cigarette alternatives
Reduced smoking | 14 days following intake date, as well as 1 month and 6 months after intake date
  Whether subjects report reduced smoking will be used to measure reduced smoking habits

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ayres, PhD, Principal Investigator — Yale Law School; Giuseppe Mattiacci, PhD, Principal Investigator — University of Amsterdam
Locations (2):
- General New Haven Public, New Haven, Connecticut, United States
- Ukraine site, Kiev, Ukraine